CLINICAL TRIAL: NCT06518200
Title: ATOPE-PRO: Effects on the Prevention of Breast Cancer Therapy-related Cardiovascular Toxicity of a Daily-adapted and Individualized Program With Support From a Mobile Application
Brief Title: Preventing Breast Cancer Therapy-related Cardiovascular Toxicity With a Daily-adapted Program With Mhealth Support
Acronym: ATOPE-PRO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Hospital Clinico Universitario San Cecilio (Other)
Responsible Party: Principal Investigator, Irene Cantarero Villanueva, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PI23/01646
Record Dates: First submitted 2024-07-11; First posted 2024-07-24 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Female
Keywords: Breast Neoplasms; Cancer therapy-related cardiovascular toxicity; Physical Exercise; Prevention; Quality of life; Rehabilitation; Telemedicine; Health related lifestyle
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double masking until end of intervention and evaluations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Individualised health recommendations + Individualised exercise intervention
  Interventions: Behavioral: Individualised health recommentations; Behavioral: Individualised physical exercise program
- Control Group (Other): General health recommendations
  Interventions: Behavioral: General health recommendations

INTERVENTIONS:
Behavioral: Individualised health recommentations — Individualised recommendations for physical activity and exercise, lifestyle, stress management and symptom management with solid scientific evidence established by health organisations and scientific reference committeess through the ATOPE-PRO mobile application based on patients reported status.
  Arms: Intervention Group
Behavioral: General health recommendations — Recommendations for physical activity and exercise, lifestyle, stress management and symptom management with solid scientific evidence established by health organisations and scientific reference committeess through the ATOPE-PRO mobile application.
  Arms: Control Group
Behavioral: Individualised physical exercise program — Follow-up of an individualised exercise program adjusted by daily monitoring of the level of physical, physiological and psychological condition.
  Arms: Intervention Group

SUMMARY:
ATOPE-PRO, was developed with the intention of consolidating the integration of an innovative system for the prevention of cancer therapy-related cardiovascular toxicity (CTR-CVT) in the continuum care of women with breast cancer in health services. It is a step further towards personalized medicine by optimizing the already available tools and integrating artificial intelligence. Breast cancer survival increases every year, a situation that poses new challenges for health professionals. The European Society for Medical Oncology, a reference in Europe, has just highlighted the need to anticipate to and prevent sequelae derived from the disease and its treatments. This, in addition to having a positive impact on improving the quality of life of people suffering from this disease, would mean a reduction in the risk of recurrence, the appearance of other tumors and other diseases, and death from cancer or other causes, which have a personal impact and represent an overload of the healthcare system. To this end, ATOPE- PRO aims to optimize and refine tools already developed in the previous project (ATOPE, Pl18/01840), integrating artificial intelligence to help identify CTR-CVT, risk profiles, and effective and safe doses (at a clinical level) early on, implementing the program in a longer term, and transferring the results to the social sector (social level). The project has 4 stages: Phase 0 or start-up (to make improvements and analyse usability); Phase 1 for piloting and optimization; Phase 2, to verify efficacy (randomized controlled clinical trial) and Phase 3, in which a deep analysis will be performed and future projects will be conceived.

DETAILED DESCRIPTION:
More and more women are experiencing breast cancer at younger ages, yet survival rates have become very promising. However, years after cancer treatment, related sequelae (physical, psychological, or emotional) may emerge, responsible for post-disease fatalities in many women. The occurrence of these sequelae largely depends on treatment-induced toxicity and individual health status, which is related to lifestyle habits. Among these sequelae, cancer-related cardiovascular toxicity (CTR-CVT) is noteworthy, with an incidence close to 40% in breast cancer, closely linked to treatments such as chemotherapy (especially anthracyclines), targeted therapy (trastuzumab), and radiotherapy (left side or mediastinum), causing DNA and mitochondrial damage. Traditionally defined as a reduction in left ventricular ejection fraction (LVEF) ≥50% in its mildest form, and a decrease in global longitudinal strain (GLS) of >15% from baseline and/or an increase in cardiac markers (cardiac troponin I or T cTnI/cTnT >99th percentile, brain natriuretic peptide BNP ≥35 pg/mL, or NT-proBNP ≥125 pg/mL) to severe (requiring inotropic support, mechanical circulatory support, or consideration for transplantation), adding the need for monitoring through various tests, not just LVEF, as it would be too late to detect it. The risk detection of TCVRC is based on medical treatments, which sometimes are insufficient since many patients theoretically considered low-risk develop TCVRC. This has led to the need to study and include other patient-related factors at the time of diagnosis, such as previous presence of cardiovascular diseases, age, lifestyle habits, and comorbidities, to be considered for overall cardiovascular and oncological prognosis and individualized surveillance of TCVRC, along with additional factors that add to the complexity of risk assessment such as cancer type, duration, and doses of oncological treatment. However, the scientific evidence supporting the inclusion of some of these parameters is of questionable quality (level C) and, moreover, they are not usually included in routine assessments, making them less applicable.

To improve the situation and achieve proper prevention of TCVRC, it is necessary to identify parameters with good sensitivity for early detection that can preferably be performed routinely by different healthcare professionals involved in the continuum of care, as well as related risk factors. With this information, the implementation of interventions that could limit treatment interruptions and improve survival after breast cancer would be facilitated. In this context, the European Society of Cardiology Guidelines highlight, in addition to the improvement of detection tools, the inclusion of new parameters, the creation of large data registries, the use of artificial intelligence, or the determination of new risk stratification algorithms, among others.

There is a lack of access to structured physical exercise programs for cancer patients, even though adaptation of exercise to their health status is crucial, as excessive doses could be harmful. Ondulatory exercise prescription may be more suitable for cancer patients, as it allows better adaptation to their health status. So far, one of the systems to achieve this has been prescription based on heart rate variability (HRV) previously used in the sports world and in some cardiovascular pathologies but promising and little studied in the cancer world. However, given the complexity of this disease, its treatments, and the impact it has on different spheres of these patients' health, the inclusion of additional markers is suggested to further optimize personalized exercise programs based on individual needs. With the support of current technologies, monitoring and control of physiological parameters are facilitated, potentially reducing the costs of in-person supervision by healthcare professionals but also the potential health risks in these patients when engaging in physical exercise.

Regarding these interventions, both physical activity and exercise have been recognized as potent multi-effect non-pharmacological therapies in the treatment of TCVRC, although to achieve optimal physiological adaptations and individualization, physical exercise programs must be correctly prescribed. In recent years, interest has shifted towards supervised high-intensity interval exercise, which has been shown to be safe, well-tolerated, effective for TCVRC treatment, and cost-effective. However, most physical exercise programs implemented are general programs with linear prescriptions and questionable adherence. To address adherence issues, physical exercise programs have been combined with behavioral change programs, showing promising short-term results but with loss in the medium/long term. In this regard, the use of technology and patient monitoring, which provide continuous feedback and have proven to be an effective and useful tool for establishing a healthy lifestyle, could offer a solution for both patients and professionals in improving adherence.

ATOPE-PRO aims to integrate into the usual care continuum of women with breast cancer a personalized and individualized mhealth model (ATOPE+ 2.0) for TCVRC prevention, which will allow us to advance towards precision clinical care, to complete its implementation and transfer of results, resulting in an improvement in quality of life, recurrence, and death, meeting the standards requested, through refining and automating the process, ensuring adherence, and offering safe and effective doses of physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed with stage I-III breast cancer
* Treatments predisposing to cardiotoxicity (anthracyclines, targeted therapies, radiotherapy)
* Signed informed consent form
* Medical authorisation to participate
* Smartphone user level

Exclusion Criteria:

* Patient underwent previous cancer treatments.
* Patients were previously diagnosed with cancer
* Pregnant patients. Patients performing other type of therapeutic exercise at diagnosis time with an intake >or = to 150 moderate-intensity or 75 min of vigorous-intensity a day
* Therapeutic exercise practice not recommended because psychiatric or cognitive disorders or cute or chronic condition that prevents exercise (advanced lung disease, oxygen requirement, stenosis >70%, metastasis etc.).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiotoxicity | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Echocardiography: left ventricular ejection fraction expressed as percentage.
Systolic function | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Echocardiography: Strain longitudinal global expressed as percentage.

SECONDARY OUTCOMES:
Number of cardiovascular events | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Clinical records registration expressed as number (N) of cardiovascular events.
Comorbidities | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Any chronic pathological condition different from the oncologic one will be registed by a clinical interview, an expressed in results as number (N) and type.
Heart rate variability | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Assessment of cardiac autonomic system balance by a Holter registration, registering the log-transformed root mean square of successive R-R intervals (lnRMSSD) and expressed as milliseconds (ms).
Heart rate | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Resting heart rate registration by a Holter, expressed as beats per minute (bpm).
Blood pressure | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Systolic and diastolic blood pressure levels registration after evaluation by a digital sphygmomanometer, expressed as mmHg (mercury millimetres).
Cardiac damage | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Collection of capillary samples for Cardiac troponin T measurement, with results expressed as ng/L, indicating higher values thatn 40ng/L cardiotoxicity or other cardiac injuries.
Cardiac Damage | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Blood test for high-sensitivity cardiac troponin I evaluation, considering normal values below 14ng/L.
Endothelial status | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  By registering ascorbic acid levels provided by blood test, being the reference range of 0.6-2 mg/dL
Cardiorespiratory Fitness | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  A Treadmill Ergometric Test will be performed in order to evaluate VO2 peak values, calcultated as the highest VO2 value in liters per minute during the test. Cut-off points will be set at low(<13 mL·kg-1·min-1), moderate (13.916.9 mL·kg-1·min-1), and high (≥17 mL·kg-1·min-1), considering a minimal clinically important difference a 6% of Vo2 peak change.
Quadriceps muscle thickness | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Quadriceps muscular ecography will be used, expressing results as centimeters (cm).
Body Fat Mass | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Bioelectrical impedance analysis (BIA) will be perfomerd by using an Inbody 720 for measuring body fat mass, expressed in kilograms (kg).
Height | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Bioelectrical impedance analysis (BIA) will be perfomerd by using an Inbody 720 for measuring body fat mass, expressed in kilograms (kg).
  A tallimeter will be used to register height, expressed in meters (m).
Weight | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Bioelectrical impedance analysis (BIA) will be perfomerd by using an Inbody 720 for measuring body weight, expressed in kilograms (kg).
Body Mass Index | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  By registering height and weight, Body mass index (BMI) will be calculated as weight (kg)/ height (m^2), expressed as kg/m^2.
Body Fat Percentage | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Bioelectrical impedance analysis (BIA) will be perfomerd by using an Inbody 720 for measuring body fat percentage, expressed as a percentage (%).
Physical Activity level | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  International physical activity questionnaire (IPAQ) will be used to report physical activity levels of participants, expressed as Metabolic Equivalent of Task per week (METs/week).
Sleep duration | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Sleep duration time, expressed as hours (h), will be recorded by activity bracelets.
Fatigue | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  A Likert 0-10 scale will be applied, indicating 0 the absence of the symptom, and a 10 'the most' of the symptom.
Total Cholesterol | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Total cholesterol (TC) will be obtained through blood test and expressed as mg/dl.
Triglycerides level | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Obtained through blood test and expressed as mmol/L.
LDL-C level | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Low-density lipoprotein cholesterol will be obtained through blood test and expressed as mg/dl.
HDL-C level | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  High-density lipoprotein cholesterol will be obtained through blood test and expressed as mg/dl.
Total antioxidant capacity | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Oxidative Stress TAC biomarker will be assessed by blood test, expressing its results as mM-TE units.
Oxidative status | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Thiobarbituric Acid Reactive Substances concentration Oxidative Stress TBARS biomarker will be assessed by blood test, being results expressed as the number of milligrammes of malonaldehyde per kilogramme of sample
Epigenetic profile | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  miRNA expression profile quantification: analysis of miRNA expression profile by massive sequencing with specific equipment, reporting changes in expression pre and post intervention as Log2 fold change (Log2FC).
Inflammatory status | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  C-reactive protein levels obtained by blood samples, expressed as mg/dl.
Immune status | At diagnosis before treatments, after 6 months, and one year after diagnosis.
  Interleuquin-6 (IL-6) levels obtained by blood samples, expressed as pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cantarero Villanueva, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Postigo-Martin P, Penafiel-Burkhardt R, Gallart-Aragon T, Alcaide-Lucena M, Artacho-Cordon F, Galiano-Castillo N, Fernandez-Lao C, Martin-Martin L, Lozano-Lozano M, Ruiz-Vozmediano J, Moreno-Gutierrez S, Illescas-Montes R, Arroyo-Morales M, Cantarero-Villanueva I. Attenuating Treatment-Related Cardiotoxicity in Women Recently Diagnosed With Breast Cancer via a Tailored Therapeutic Exercise Program: Protocol of the ATOPE Trial. Phys Ther. 2021 Mar 3;101(3):pzab014. doi: 10.1093/ptj/pzab014. PMID 33528004
- [Background] Gonzalez-Santos A, Postigo-Martin P, Gallart-Aragon T, Esteban-Cornejo I, Lopez-Garzon M, Galiano-Castillo N, Arroyo-Morales M, Illescas-Montes R, Artacho-Cordon F, Martin-Martin L, Forneiro-Perez R, Lozano-Lozano M, Fernandez-Lao C, Ruiz-Vozmediano J, Sanchez-Salgado C, Cantarero-Villanueva I. Neurotoxicity prevention with a multimodal program (ATENTO) prior to cancer treatment versus throughout cancer treatment in women newly diagnosed for breast cancer: Protocol for a randomized clinical trial. Res Nurs Health. 2021 Aug;44(4):598-607. doi: 10.1002/nur.22136. Epub 2021 May 7. PMID 33963594
- [Result] Postigo-Martin P, Gil-Gutierrez R, Moreno-Gutierrez S, Lopez-Garzon M, Gonzalez-Santos A, Arroyo-Morales M, Cantarero-Villanueva I. mHealth system (ATOPE+) to support exercise prescription in breast cancer survivors: a reliability and validity, cross-sectional observational study (ATOPE study). Sci Rep. 2022 Sep 8;12(1):15217. doi: 10.1038/s41598-022-18706-7. PMID 36076044
- [Result] Gonzalez-Santos A, Lopez-Garzon M, Gil-Gutierrez R, Salinas-Asensio MDM, Postigo-Martin P, Cantarero-Villanueva I. Nonlinear, Multicomponent Physical Exercise With Heart Rate Variability-Guided Prescription in Women With Breast Cancer During Treatment: Feasibility and Preliminary Results (ATOPE Study). Phys Ther. 2023 Sep 1;103(9):pzad070. doi: 10.1093/ptj/pzad070. PMID 37347987
- See also: S. Moreno-Gutierrez et al., "ATOPE+: An mHealth System to Support Personalized Therapeutic Exercise Interventions in Patients With Cancer," in IEEE Access, vol. 9, pp. 16878-16898, 2021, doi: 10.1109/ACCESS.2021.3049398. — https://ieeexplore.ieee.org/document/9314150